CLINICAL TRIAL: NCT05199142
Title: A Phase 1b, Exploratory, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of SDI-118 in Elderly Male and Female Study Participants With Cognitive Decline
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of SDI-118 in Elderly Male and Female Study Participants With Cognitive Decline
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development plan changed
Sponsor: Syndesi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYND005
Record Dates: First submitted 2021-11-30; First posted 2022-01-20 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDI-118 (Experimental): SDI-118 capsule self-administered orally once daily (QD) for 17 days.
  Interventions: Drug: SDI-118
- Placebo (Placebo Comparator): Placebo capsule self-administered orally once daily (QD) for 17 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SDI-118 — SDI-118 Powder in Capsules (PiC) are presented as Drug Substance in white, size 3, hydroxypropylmethylcellulose (HPMC) capsules. No excipients are added.
  Arms: SDI-118
Drug: Placebo — The Matching Placebo for SDI-118 PiC is equivalent dose of mannitol (an inert excipient) in white, size 3, hydroxypropylmethylcellulose (HPMC) capsules.
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, randomized, placebo-controlled study to determine the safety, tolerability, and pharmacodynamics of SDI-118 in a once daily (QD) dosing regimen on elderly male and female study participants with cognitive decline at screening.

ELIGIBILITY:
Inclusion Criteria:

* Male and female study participants between 65 and 85 years of age (inclusive) at screening, with cognitive decline, defined as:

  * >25 on the MMSE;
  * <11 on the GDS; and
  * IQCODE score of ≥52.
* Participants with delayed recall of ≤6 words from the ISLT 15 minutes after the presentation of the word list;
* Must be in good health for their age as determined by medical history, physical examinations, 12-lead ECGs, vital signs, and clinical laboratory assessments (serum chemistry, serum hematology, and urinalysis) performed at the Screening Visit;
* Must have an informant (eg, spouse, family member, caregiver, or other close contact) who has known the study participant for at least 10 years to provide data on the study participant;
* Negative serology tests for HIV antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies at screening;
* Have a body mass index of 18 to 36 kg/m2 inclusive;
* Agree not to use herbal medications (including herbal tea, St. John's Wort), within 14 days prior to study drug administration to the Safety Follow-Up Visit (Visit 7);
* Agree not to use previously prescribed medications that are expected to interfere with the absorption, distribution, metabolism, and/or excretion (ie, strong cytochrome P450 3A4 or 2C19 inhibitors or inducers, LEV, and brivaracetam) or safety/tolerability evaluation of SDI-118 or that could interfere with the objectives of the study (ie, medications with CNS activity);
* Participants must have signed an informed consent document indicating that the participants understand the purpose of, and procedures required for the study, and are willing to participate in the study;
* Smokers are allowed if their average daily consumption does not exceed 5 cigarettes per day (or maximum equivalent of 5 cigarettes per day);
* Non-vasectomized male participants with a female partner of childbearing potential must agree to use a condom from first dosing up to 90 days after the last dose. Additionally, the female partner must be willing to use a highly effective method of contraception;
* Female participants must have confirmed menopause;
* The participant, in the opinion of the Investigator, is willing and able to adhere to the study visit schedule and other requirements, prohibitions, and restrictions of the study.

Exclusion Criteria:

* Are left-handed;
* Have, or have a history within the last 12 months of, drug or alcohol dependency or positive urine drug screen or alcohol breath test at Screening or Assessment Visits;
* History, or presence upon clinical examination, of cardiac, ophthalmologic, pulmonary, endocrine (uncontrolled diabetes), cancer, blood disease, gastrointestinal, hepatic, renal disease, or other condition that, in the opinion of the Investigator, could interfere with the test procedures;
* History or presence of significant neurological or psychiatric conditions such as stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, or blackouts requiring hospitalization;
* History of, or current condition of, migraine headaches;
* Have undergone operations to the brain;
* Have significant visual impairment including color blindness, history of ocular treatment including corrective laser eye surgery, or ongoing condition that, in the opinion of the Investigator, may interfere with the performance of the cognitive test battery;
* Participants who consume large amounts of caffeinated drinks (more than 8 cups of standard caffeinated drinks [eg, tea, instant coffee] or 6 cups of stronger coffee or other drinks containing methylxanthines such as soda or energy drinks per day);
* Have received an experimental drug and/or used an experimental medical device within 30 days of the Screening Visit or within 5 half-lives, whichever is longer;
* Are unable to comply with MRI Patient Declaration;
* Have a resting pulse <45 bpm or >100 bpm at Screening or on Day 1;
* Participants with any of the following findings in the resting ECG:

  * Fridericia-corrected QT interval >450 ms (males); >470 ms (females); or <300 ms at Screening or on Day 1; or
  * Wolff-Parkinson-White syndrome, complete left bundle branch block (LBBB).
* Family history of congenital long QT syndrome or sudden death;
* Poorly controlled diabetes (hemoglobin A1c >8.5%);
* Poorly controlled hypertension (systolic blood pressure >155 mmHg and diastolic blood pressure >95 mmHg);
* Diagnosed with anemia (defined as hemoglobin <12 g/dL);
* Have reduced renal function defined as having an estimated glomerular filtration rate (eGFR) of <59 mL/min/1.73 m²;
* Have physical, language, or other impairments of such severity as to adversely affect the validity of the data derived from the cognitive tasks as judged by the Investigator;
* Any suicidal ideation of type 4 or 5 in the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past 3 months prior to screening or at Screening or Baseline Visits;
* Unable to comply with MRI or blood draw procedures (suffers from claustrophobia or needle phobia);
* Known clinically relevant structural brain abnormality as determined by previous MRI or persistent MRI imaging artefact which is judged to produce extensive imaging distortions (eg, extensive dental work) as determined at the Imaging Baseline Visit (Visit 2, Day 0); or
* With a disease or take any medication that, in the Investigator's and/or Sponsor's opinion, could interfere with the assessments of safety, tolerability, or pharmacodynamics as well as the conduct or interpretation of the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 17 days
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered a study drug and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical product whether or not considered related to the medical product. An AE is considered "serious" if, in the view of either the investigator or sponsor, the event: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires hospitalization or prolongation to hospitalization, or other medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | 17 days
  Number of participants with potentially clinically significant laboratory values (hematology/chemistry/urinalysis).
Number of participants with vital sign abnormalities and/or adverse events (AEs) | 17 days
  Number of participants with potentially clinically significant vital sign values.
Number of participants with routine 12 lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant ECG values.
Number of participants with C-SSRS abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in C-SSRS values.
Number of participants with routine physical examination abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in physical examination.
Number of participants with Changes in the Cogstate Brief Battery, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the Cogstate Brief Battery values.
Number of participants with Changes in the Digital Symbol Substitution Test, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the DSST values.
Number of participants with Changes in the Controlled Oral Word Association Test, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the COWAT values.
Number of participants with Changes in the Category Fluency Test, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the CFT values.

SECONDARY OUTCOMES:
Changes in Blood Oxygen Level Dependent (BOLD) signal | 17 days
  As measured by changes in deoxyhemoglobin levels driven by localized changes in brain blood flow and blood oxygenation in brain networks associated with executive function (working memory), including the prefrontal cortex, the hippocampus, and the associated limbic networks, during performance of the N-Back Tasks
Performance measures associated with executive function (working memory) during the N-Back Tasks | 17 days
  As measured by both response accuracy and response latency between cue stimulus and detection of this cue in the presented trial stimuli

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Frankfurt, Frankfurt am Main, Germany
- St Pancras Clinical Research, London, United Kingdom